CLINICAL TRIAL: NCT03725007
Title: An Open-Label Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Upadacitinib in Pediatric Subjects With Polyarticular Course Juvenile Idiopathic Arthritis
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Upadacitinib in Pediatric Subjects With Polyarticular Course Juvenile Idiopathic Arthritis
Acronym: SELECT-YOUTH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M15-340; 2018-000715-25 (EudraCT Number)
Record Dates: First submitted 2018-10-27; First posted 2018-10-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: Upadacitinib; ABT-494; Polyarticular Course Juvenile Idiopathic Arthritis (pcJIA)
MeSH Terms: conditions — Arthritis, Juvenile | interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Participants of age group 12 to <18 years receiving dose A (Experimental): Participants of age group 12 to <18 years administered with upadacitinib dose A (weight dependent) as described in the protocol.
  Interventions: Drug: Upadacitinib
- Participants of age group 12 to <18 years receiving dose B (Experimental): Participants of age group 12 to <18 years administered with upadacitinib dose B (weight dependent) as described in the protocol.
  Interventions: Drug: Upadacitinib
- Participants of age group 6 to <12 years receiving dose A (Experimental): Participants of age group 6 to <12 years administered with upadacitinib dose A (weight dependent) as described in the protocol.
  Interventions: Drug: Upadacitinib
- Participants of age group 2 to <6 years receiving dose A (Experimental): Participants of age group 2 to <6 years administered with upadacitinib dose A (weight dependent) as described in the protocol.
  Interventions: Drug: Upadacitinib
- Participants of age group 2 to <18 years receiving dose A (Experimental): Participants of age group 2 to <18 years administered with upadacitinib dose A as described in the protocol.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib is administered as an oral solution or tablet as described in protocol.
  Other Names: ABT-494

SUMMARY:
This is a study to evaluate pharmacokinetics, safety and tolerability of upadacitinib in pediatric participants with polyarticular course juvenile idiopathic arthritis. This study consists of three parts: Part 1 is multiple-cohort study that consists of two sequential multiple dose groups. Participants benefiting from the study drug with no ongoing adverse events of special interest or serious adverse events will have option to enroll in Part 2. Part 2 is open-label, long term extension study to evaluate safety and tolerability. Part 3 is an additional safety cohort to evaluate long-term safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Participant have total body weight of 10 kg or higher at the time of screening.
* Participant diagnosed with pcJIA (rheumatoid factor-positive or rheumatoid factor-negative polyarticular JIA, extended oligoarticular JIA, or systemic JIA with active arthritis and without active systemic features) with a history of arthritis affecting at least 5 joints within the first 6 months of disease (for extended oligoarticular JIA: <=4 joints within first 6 months of disease and >4 joints thereafter).
* Participant have 5 or more active joints at the time of screening, defined as the presence of swollen joints (not due to deformity) or, in the absence of swelling, joints with the limitation of movement (LOM) plus pain on motion and/or tenderness with palpitation, with LOM present in at least three of the active joints.
* If receiving methotrexate (MTX), have been taking MTX for at least 12 weeks immediately before and including Study Day 1 on a stable dose of <=20 mg/m2 for at least 8 weeks before and including Study Day 1; in addition, participants should take either folic acid or folinic acid according to local standard of care.
* If on oral glucocorticosteroids, must have been taking oral glucocorticosteroids at a stable dose (no greater than 10 mg/day or 0.2 mg/kg/day, whatever is lower) for at least 1 week before and including Study Day 1.

Exclusion Criteria:

* Participant with diagnosis of enthesitis-related arthritis (ERA) or juvenile psoriatic arthritis (JPSA).
* Participant have prior exposure to JAK inhibitor.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | Up to approximately 156 weeks
  Adverse Event is defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product.
Part 1: Maximum observed plasma concentration (Cmax) | Day 7
  Cmax is defined as the maximum observed plasma concentration for upadacitinib.
Part 1: Time to maximum observed plasma concentration (Tmax) | Day 7
  Tmax is defined as the time to maximum plasma concentration (Cmax) of upadacitinib.
Part 1: Area under plasma concentration versus time curve during a dosing interval (AUCtau) | Day 7
  The area under the plasma concentration-time curve is a method of measurement of the total exposure of a drug in plasma.
Part 1: Apparent oral clearance at steady state (CL/F) | Day 7
  Clearance is defined as the volume of plasma cleared of the drug per unit time.
Part 1: Half-life | Day 7
  Half life of updadacitinib will be determined using non-compartmental method.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (35):
- United States (8):
  - Ann & Robert H Lurie Children's Hospital of Chicago /ID# 211162, Chicago, Illinois
  - Duplicate_University of Louisville /ID# 202896, Louisville, Kentucky
  - Boston Children's Hospital /ID# 202993, Boston, Massachusetts
  - Cincinnati Childrens Hospital Medical Center /ID# 209697, Cincinnati, Ohio
  - Randall Children's Hospital /ID# 213609, Portland, Oregon
  - Children's Hospital of Philadelphia /ID# 209617, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC /ID# 202994, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital /ID# 203003, Seattle, Washington
- Canada (3):
  - Alberta Children's Hospital /ID# 251738, Calgary, Alberta
  - British Columbia Children and Women's Hospital and Health Centre /ID# 251736, Vancouver, British Columbia
  - Duplicate_McGill University Health Centre /ID# 251252, Montreal, Quebec
- Germany (5):
  - Asklepios Klinik Sankt Augustin /ID# 203264, Sankt Augustin, North Rhine-Westphalia
  - St. Josef-Stift Sendenhorst /ID# 244740, Sendenhorst, North Rhine-Westphalia
  - PRI - Pediatric Rheumatology Research Institute /ID# 205954, Bad Bramstedt, Schleswig-Holstein
  - Helios Klinikum Berlin-Buch /ID# 206859, Berlin
  - Hamburger Zentrum fuer Kinder- und Jugendrheumatologie /ID# 206571, Hamburg
- Semmelweis Egyetem /ID# 208970, Budapest, Hungary
- The Chaim Sheba Medical Center /ID# 222370, Ramat Gan, Tel Aviv, Israel
- Ospedale Pediatrico Bambino Gesù /ID# 203835, Rome, Roma, Italy
- Japan (7):
  - Aichi Children's Health and Medical Center /ID# 248327, Obu-shi, Aichi-ken
  - Hyogo Prefectural Kobe Children's Hospital /ID# 246582, Kobe, Hyōgo
  - Kagoshima University Hospital /ID# 246501, Kagoshima, Kagoshima-ken
  - St Marianna University School Of Medicine /ID# 246478, Kawasaki-shi, Kanagawa
  - Miyagi Children's Hospital /ID# 246734, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital /ID# 247246, Niigata, Niigata
  - Institute of Science Tokyo Hospital /ID# 246500, Bunkyo-ku, Tokyo
- Puerto Rico (3):
  - Centro de Reumatologia Pediatrico de Puerto Rico /Id# 204406, Bayamón
  - GCM Medical Group PSC /ID# 211702, San Juan
  - Mindful Medical Research /ID# 204488, San Juan
- Spain (5):
  - Hospital Sant Joan de Deu /ID# 203915, Esplugues de Llobregat, Barcelona
  - Hospital Infantil Universitario Nino Jesus /ID# 206466, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 203917, Madrid
  - Hospital Universitario La Paz /ID# 203927, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 203914, Valencia
- Queen Silvia Children's Hosp /ID# 251145, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No